CLINICAL TRIAL: NCT05857722
Title: Improving Mental Health Among Colombian and Venezuelan Youth Affected by Forced Displacement
Acronym: JC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Brown University (Other); Universidad de Los Andes (Unknown)
Responsible Party: Principal Investigator, Maria Pineros Leano, Assistant Professor, Boston College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27332
Record Dates: First submitted 2023-04-21; First posted 2023-05-15 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Emotion Regulation; Mood Disorders
Keywords: Intervention; Implementation; Venezuelan migrants; Internally displaced population; Forced migration; Mental health; Emotion regulation
MeSH Terms: conditions — Emotional Regulation; Mood Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will recruit and enroll 120 male/120 female youth (N=240) aged 18-30 from several communities in Bogotá using stratified selection for gender balance; and then randomize youth to receive Jóvenes Capibara within entrepreneurship training (N=120) or to a waitlist condition (N=120). Waitlisted youth will be eligible to receive the intervention after 6-month follow-up data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entrepreneurship and Jóvenes Capibara group (Experimental): Participants in the experimental arm will receive a 10-day intervention, which consists of an entrepreneurship program, plus Jóvenes Capibara, an intervention that aims to improve emotion regulation and mental health symptoms among youth impacted by violence.
  Interventions: Behavioral: Jóvenes Capibara
- Control waitlist condition (Other): Participants in the control waitlist condition will will be eligible to receive the intervention after 6-month follow-up data collection, which will take place approximately 10 to 12 months after the Entrepreneurship and Jóvenes Capibara group receives the intervention.
  Interventions: Behavioral: Jóvenes Capibara

INTERVENTIONS:
Behavioral: Jóvenes Capibara — Jóvenes Capibara is a 10-session group intervention that was culturally adapted from the Youth Readiness Intervention, which was originally developed in Sierra Leone for conflict-affected youth. Jóvenes Capibara was adapted to the Colombian context using the ADAPT-ITT framework, which ensured that the intervention was relevant to the needs of Colombian and Venezuelan youth.
  Other Names: Youth Readiness Intervention

SUMMARY:
The goal of this randomized controlled trial is to test the effectiveness of an emotion regulation intervention called Jóvenes Capibara in a Venezuelan migrant and internally displaced population sample of youth between the ages of 18 through 30 delivered within a 10-day boot-camp entrepreneurship program. The main questions it aims to answer are: (a) Is Jóvenes Capibara feasible and acceptable among internally displaced population and Venezuelan migrant youth aged 18-30 in Colombia?; (b) Is delivery of Jóvenes Capibara within entrepreneurship training feasible and acceptable among facilitators?; (c) Is Jóvenes Capibara associated with improved mental health, daily functioning, and labor market outcomes in Colombian and Venezuelan youth who receive the intervention compared with youth in the control group? Participants will receive a 10-day intervention, which consists of an entrepreneurship program, plus Jóvenes Capibara, an intervention that aims to improve emotion regulation and mental health symptoms among youth impacted by violence. Measures will be taken at baseline, post-intervention, and at 6-month post-intervention follow-up. The comparison group will receive the intervention one year after youth in the experimental condition. The researchers will compare the experimental group and the waitlist control group to determine the effects of Jóvenes Capibara on mental health, daily functioning, and labor market outcomes.

DETAILED DESCRIPTION:
The investigators will recruit and enroll 120 male/120 female youth (N=240) aged 18-30 from several communities in Bogotá using stratified selection for gender balance; and then randomize youth to receive Jóvenes Capibara within entrepreneurship training (N=120) or to a waitlist condition (N=120). Waitlisted youth will be eligible to receive the intervention after 6-month follow-up data collection. A codified set of randomization rules will minimize contamination risks, and a computer-generated randomization allocation sequence will guide randomization procedures.

Measures, Data Points, and Data Analysis Strategy: The investigators will collect quantitative data on mental health and daily functioning at baseline, post-intervention, and 6-month follow-up. The investigators will collect qualitative and quantitative data at post-intervention from facilitators on implementation outcomes (feasibility, acceptability, adoption, appropriateness). The investigators will use the Difficulties in Emotion Regulation Scale (DERS), General Self-Efficacy Scale, WHO Disability Assessment Schedule (WHODAS), Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder Screener (GAD-7), PTSD Checklist-Civilian Version (PCL-C), and the Demographic and Household Scale IPV items (DHS-IPV). The investigators will also assess labor market outcomes, including employment, hours worked, and income earned at each time point. A subset of youth (n=24) selected based on a multivariate sampling matrix will complete exit interviews to assess feasibility, acceptability and satisfaction with the intervention.

The investigators will use mixed linear effects modeling to investigate the clinical effectiveness of the Jóvenes Capibara on mental and behavioral health outcomes among youth. The investigators will compare Jóvenes Capibara participants to those in the control condition to assess whether there is significantly greater change in mental health, emotion regulation, daily functioning, and labor market outcomes over time among Jóvenes Capibara participants. The investigators will use mixed effects linear models to assess the impact of the intervention on quantitative mental health outcomes. These models will account for clustering of individual outcomes among lay health workers delivering the Jóvenes Capibara as well clustering of outcomes within individuals across time points. In cases where the outcome scale scores are skewed and violate the normality assumption for linear models, the investigators will use generalized linear models with a Poisson distribution. The investigators will include a time dummy variable to account for time effects and treatment by time interaction terms to test the impact of the treatment on outcomes at post-intervention and 6-month follow-up. All analyses will be conducted on an intent-to-treat basis.

Power considerations will assess our primary hypothesis -Jóvenes Capibara youth will report significantly greater mental health benefits than control youth. The investigators assume a standardized mean difference between intervention and control conditions of approximately 0.30-0.45 to determine Jóvenes Capibara effectiveness on youth mental health outcomes, which corresponds to the effect sizes observed in our prior studies. Assuming a standard alpha level of <0.05 with data from 2 time points with a moderate intra-class (within individual) correlation of approximately 0.5, and accounting for 20% attrition, this RCT has power of 0.80 to detect a standardized medium effect size of approximately 0.35.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 18-30
* Venezuelan migrant or Colombian who has been internally displaced or directly/indirectly impacted by internal conflict in Colombia

Exclusion Criteria:

* Current suicidality or homicidality
* Psychosis
* Serious medical condition, or severe cognitive impairment that would preclude ability to participate in study assessments and activities, as assessed via the MINI-SCID by a study psychologist.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 296 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | Baseline
  18-item scale that measures emotion regulation using a 1-5 Likert scale. Lower scores indicate worse emotion regulation.
Difficulties in Emotion Regulation Scale (DERS) | Immediately post-intervention
  18-item scale that measures emotion regulation using a 1-5 Likert scale. Lower scores indicate worse emotion regulation.
Difficulties in Emotion Regulation Scale (DERS) | 6 month follow-up: up to 8 months post-baseline
  18-item scale that measures emotion regulation using a 1-5 Likert scale. Lower scores indicate worse emotion regulation.
World Health Organization Disability Assessment Schedule (WHODAS) | Baseline
  36-item scale that measures self-rated disability using a 5 point Likert scale ranging from 1 (none) to 5 (extremely or cannot do it). Higher scores indicate higher levels of disability.
World Health Organization Disability Assessment Schedule (WHODAS) | Immediately post-intervention
  36-item scale that measures self-rated disability using a 5 point Likert scale ranging from 1 (none) to 5 (extremely or cannot do it). Higher scores indicate higher levels of disability.
World Health Organization Disability Assessment Schedule (WHODAS) | 6 month follow-up: up to 8 months post-baseline
  36-item scale that measures self-rated disability using a 1-5 point Likert scale ranging from 1 (none) to 5 (extremely or cannot do it). Higher scores indicate higher levels of disability.
Patient Health Questionnaire (PHQ-9) | Baseline
  9-item depression scale. This scale uses a 0-3 Likert scale. Lower levels indicate fewer symptoms of depression.
Patient Health Questionnaire (PHQ-9) | Immediately post-intervention
  9-item depression scale. This scale uses a 0-3 Likert scale. Lower levels indicate fewer symptoms of depression.
Patient Health Questionnaire (PHQ-9) | 6 month follow-up: up to 8 months post-baseline
  9-item depression scale. This scale uses a 0-3 Likert scale. Lower levels indicate fewer symptoms of depression.
Generalized Anxiety Disorder Screener (GAD-7) | Baseline
  7-item anxiety scale. This scale uses a 0-3 Likert scale, with 0 being "not at all", and 3 being "nearly every day". Lower levels indicate fewer symptoms of anxiety.
Generalized Anxiety Disorder Screener (GAD-7) | Immediately post-intervention
  7-item anxiety scale. This scale uses a 0-3 Likert scale, with 0 being "not at all", and 3 being "nearly every day". Lower levels indicate fewer symptoms of anxiety.
Generalized Anxiety Disorder Screener (GAD-7) | 6 month follow-up: up to 8 months post-baseline
  7-item anxiety scale. This scale uses a 0-3 Likert scale, with 0 being "not at all", and 3 being "nearly every day". Lower levels indicate fewer symptoms of anxiety.
Post-traumatic stress disorder Checklist-Civilian Version (PTSD CL) | Baseline
  17-item post-traumatic stress scale. This scale uses a 1-5 Likert scale, with 1 being "Not at all" and 5 being "Extremely". Lower scores indicate fewer symptoms of post-traumatic stress.
Post-traumatic stress disorder Checklist-Civilian Version (PTSD CL) | Immediately post-intervention
  17-item post-traumatic stress scale. This scale uses a 1-5 Likert scale, with 1 being "Not at all" and 5 being "Extremely". Lower scores indicate fewer symptoms of post-traumatic stress.
Post-traumatic stress disorder Checklist-Civilian Version (PTSD CL) | 6 month follow-up: up to 8 months post-baseline
  17-item post-traumatic stress scale. This scale uses a 1-5 Likert scale, with 1 being "Not at all" and 5 being "Extremely". Lower scores indicate fewer symptoms of post-traumatic stress.
General Self-Efficacy Scale | Baseline
  10-item self-efficacy scale. This scale uses a 1-4 Liker scale, with 1 being "Not at all true", and 4 being "Exactly true". Lower scores indicate lower levels of self-efficacy.
General Self-Efficacy Scale | Immediately post-intervention
  10-item self-efficacy scale. This scale uses a 1-4 Liker scale, with 1 being "Not at all true", and 4 being "Exactly true". Lower scores indicate lower levels of self-efficacy.
General Self-Efficacy Scale | 6 month follow-up: up to 8 months post-baseline
  10-item self-efficacy scale. This scale uses a 1-4 Liker scale, with 1 being "Not at all true", and 4 being "Exactly true". Lower scores indicate lower levels of self-efficacy.
Demographic and Household Scale Intimate Partner Violence (DHS-IPV) | Baseline
  19-36 item questionnaire. The number of items asked depends on the number of questions endorsed. The answers are Yes [1] or No [0]. The first 5 questions are asked to everyone and they do not have skip patterns. Questions 6-35 are asked and if the answer is yes, a follow-up question is asked; otherwise, the question follow-up question is skipped. Lower levels indicate lower levels of intimate partner violence
Demographic and Household Scale Intimate Partner Violence (DHS-IPV) | Immediately post-intervention
  19-36 item questionnaire. The number of items asked depends on the number of questions endorsed. The answers are Yes [1] or No [0]. The first 5 questions are asked to everyone and they do not have skip patterns. Questions 6-35 are asked and if the answer is yes, a follow-up question is asked; otherwise, the question follow-up question is skipped. Lower levels indicate lower levels of intimate partner violence
Demographic and Household Scale Intimate Partner Violence (DHS-IPV) | 6 month follow-up: up to 8 months post-baseline
  19-36 item questionnaire. The number of items asked depends on the number of questions endorsed. The answers are Yes [1] or No [0]. The first 5 questions are asked to everyone and they do not have skip patterns. Questions 6-35 are asked and if the answer is yes, a follow-up question is asked; otherwise, the question follow-up question is skipped. Lower levels indicate lower levels of intimate partner violence
Labor market outcomes | Baseline
  Labor market outcomes are measured using a validated scale developed in Colombia. It consists of 21 questions. Questions 1-4 are Yes [1], No [2] questions. If Yes is answered on these questions, then questions 5-19 are asked. Otherwise, questions 5-19 are skipped and asked questions 20 and 21. This questionnaire asks about type of employment, number of hours worked, number of days worked within the past month, occupation, and income.
Labor market outcomes | Immediately post-intervention
  Labor market outcomes are measured using a validated scale developed in Colombia. It consists of 21 questions. Questions 1-4 are Yes [1], No [2] questions. If Yes is answered on these questions, then questions 5-19 are asked. Otherwise, questions 5-19 are skipped and asked questions 20 and 21. This questionnaire asks about type of employment, number of hours worked, number of days worked within the past month, occupation, and income.
Labor market outcomes | 6 month follow-up: up to 8 months post-baseline
  Labor market outcomes are measured using a validated scale developed in Colombia. It consists of 21 questions. Questions 1-4 are Yes [1], No [2] questions. If Yes is answered on these questions, then questions 5-19 are asked. Otherwise, questions 5-19 are skipped and asked questions 20 and 21. This questionnaire asks about type of employment, number of hours worked, number of days worked within the past month, occupation, and income.

SECONDARY OUTCOMES:
Family Care Indicators (FCI) | Baseline
  12-item questionnaire. 6 items are follow-up items to the stem question (even number questions). If the stem question is endorsed, then the follow-up question is asked. Stem question has two answers; Yes [1], No [0]. The follow-up questions ask who engaged the child on a certain activity (i.e., mother, father, other). Lower scores indicate worse child engagement outcomes.
Family Care Indicators (FCI) | Immediately post-intervention
  12-item questionnaire. 6 items are follow-up items to the stem question (even number questions). If the stem question is endorsed, then the follow-up question is asked. Stem question has two answers; Yes [1], No [0]. The follow-up questions ask who engaged the child on a certain activity (i.e., mother, father, other). Lower scores indicate worse child engagement outcomes.
Family Care Indicators (FCI) | 6 month follow-up: up to 8 months post-baseline
  12-item questionnaire. 6 items are follow-up items to the stem question (even number questions). If the stem question is endorsed, then the follow-up question is asked. Stem question has two answers; Yes [1], No [0]. The follow-up questions ask who engaged the child on a certain activity (i.e., mother, father, other). Lower scores indicate worse child engagement outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Open recruitment, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Desrosiers A, Pineros-Leano M, Saran I, Escobar C, Pineros-Leano N, Jimenez MP, Moya A, Betancourt TS. Integrating a culturally adapted mental health intervention within entrepreneurship training for displaced youth in Colombia: a pilot randomized controlled trial. Confl Health. 2025 Jul 31;19(1):54. doi: 10.1186/s13031-025-00675-z. PMID 40745658